CLINICAL TRIAL: NCT00824551
Title: The Effects of Hyperbaric Oxygen Therapy on Acute Thermal Burns
Brief Title: The Effects of Hyperbaric Oxygen Therapy (HBOT) on Acute Thermal Burns
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: chong si jack, republic of singapore navy and singapore general hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1501
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2008-12

CONDITIONS: Acute Thermal Burns
Keywords: Acute Thermal Burns; Hyperbaric Oxygen Therapy; Burns conversion
MeSH Terms: interventions — Hyperbaric Oxygenation; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperbaric Oxygen Therapy (Experimental): 2 HBOT treatments
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- 2 (Active Comparator): Standard care and treatment
  Interventions: Other: Standard care

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — 2 sessions of HBOT ( HDMC 14)
  Arms: Hyperbaric Oxygen Therapy
Other: Standard care — Patient will undergo standard care
  Arms: 2

SUMMARY:
The blinded RCTstudy aims to:

* Determine the effects of HBOT on burns conversion for patients who have fresh thermal burns injury using the LDI.
* Objectively determine the proportion of burns conversion in areas of partial thickness burns for early thermal burns injury in both arms of the RCT.
* Study the effects of HBOT on immunological markers IL-1, IL-2, IL-4, IL-6, IL-8, IL-10, TNF-α and TGF-β ( comparison between both arms and 2 assessment points).
* Study the effect of HBOT on haematological markers including procalcitonin ,albumin, lymphocyte counts, neutrophil count, and macrophage count.
* Study the effects of HBOT on histology specimens in quantifying P53 protein, leukocyte and macrophage infiltration, burns depth assessment and vascular endothelial growth factor (VEGF) and inducible nitric oxide synthase (iNOS) .
* Study the effects of HBOT on bacteriology of tissue culture in areas of deep dermal burns.

ELIGIBILITY:
Inclusion Criteria:

* Thermal burns injury less than 40% with areas of deep dermal/ full thickness burns.
* Less than 24 hours from time of injury.
* No inhalational injury (Nasoendoscopy and bronchoscopic diagnosis by burns centre medical team/ department of emergency medicine in SGH).
* Age 21 years old and above and less than 60 years old.
* Not intubated and not on inotropic support.
* Understands and agrees to informed consent (approved by IRB SGH).

Exclusion Criteria:

* Untreated pneumothorax
* Medications: Bleomycin, Cis-platin, Doxorubicin, Disulfiram (Chemotherapy)
* Acute uncontrolled medical condition or significant medical condition (eg. Cerebrovascular accident, diabetic ketoacidosis, severe hypertensive 180/ 110 mmHg, end stage renal failure, chest pain, bleeding gastrointestinal tract, coma and acute asthma attack)
* Other surgical emergencies (eg. open fractures, compartment syndrome and acute abdomen)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Burns conversion | 2 years

SECONDARY OUTCOMES:
Bacteriology culture and immunology markers | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore